CLINICAL TRIAL: NCT02008513
Title: A Randomized, Controlled, Parallel Group, Double-blind, Multi-centre, Phase IIb Study to Assess Safety and Clinical Activity of Continued AFFITOPE® AD02 Vaccinations of Patients Who Participated in the AFFITOPE® AD02 Phase II Study AFF006.
Brief Title: Follow-up Study to Assess Safety and Clinical Activity of Continued AFFITOPE® AD02 Vaccinations of Patients Who Participated in AFF006
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study AFF006A was early terminated by the sponsor based on the results of study AFF006.
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFF006A; 2012-005280-27 (EudraCT Number)
Record Dates: First submitted 2013-10-30; First posted 2013-12-11 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Alzheimer´s Disease
Keywords: AFFITOPE® AD02; Alzheimer Disease; Dementia; Brain Disease; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): AFF006 Placebo groups receive 6 AFFITOPE® AD02 vaccinations
  Interventions: Biological: AFFITOPE® AD02
- Group 2 (Active Comparator): AFF006 verum groups receive 3 Placebo injections then followed by 3 AFFITOPE® AD02 vaccinations
  Interventions: Biological: AFFITOPE® AD02; Biological: Placebo

INTERVENTIONS:
Biological: AFFITOPE® AD02
Biological: Placebo
  Arms: Group 2

SUMMARY:
This is a follow-up study to assess safety and clinical activity of continued AFFITOPE® AD02 vaccinations in patients with Alzheimer's disease. Patients, who have already participated in AFF006 will be involved in 27 study sites in Europe. Duration of patient's participation in the clinical trial is 19 months.

ELIGIBILITY:
Inclusion Criteria:

* patients having participated in AFF006+having received 6 investigational medicinal product (IMP) injections+having completed all visits
* Written informed consent
* Availability of a partner/caregiver
* Female patients of childbearing potential are eligible if they use a medically accepted contraceptive method.
* Scheduled elective hospitalization for diagnostic work-up is allowed for inclusion into the clinical trial.

Exclusion Criteria:

* Pregnant women.
* Sexually active women of childbearing potential who are not using a medically accepted birth control method and unreliable contraception in male subjects.
* Participation in the active treatment phase of another clinical trial except AFF006 within 3 months before Visit 0.
* History of questionable compliance to visit schedule; patients not expected to complete the clinical trial.
* Presence or history of allergy to components of the vaccine, if considered relevant by the investigator.
* Contraindication for MRI imaging
* Presence and/or history of immunodeficiency (e.g., HIV infection).
* Prior and/or current treatment with experimental immunotherapeutics including Intravenous immunoglobulin (IVIG), AD antibody therapy and/or vaccines for AD except AD02.
* Prior and/or current treatment with immunosuppressive drugs.
* Treatment with benzodiazepines and/or nootropics administered at high doses and/or as newly started treatment.
* Treatment with anticholinergic drugs including Parkinson treatments, antidepressants (tricyclics), neuroleptics with anticholinergic properties, certain bladder relaxants, anticholinergic drugs for use in lung diseases.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Composite Measures of Primary Safety and Tolerability Endpoints | 19 months
  * Withdrawal criteria
  * Number of Adverse events (AEs)
  * Number of any serious adverse events (SAE)
  * Alzheimer's Disease Assessment Scale - Cognition (ADAScog)
  * Alzheimer's Disease Co-operative Study - Activities of Daily Living Inventory (ADCS-ADL)

SECONDARY OUTCOMES:
Composite Measures of Secondary Efficacy Endpoints | 19 months
  * Clinical Dementia Rating Sum of Boxes (CDR-sb)
  * Free and Cued Selective Reminding Test (FCSRT)
  * Standard neuropsychological test battery (CogState)
  * Mini-Mental State Examination (MMSE)
  * Investigator's global evaluation scale (IGE)
  * CDR [global aspects]
  * Neuropsychiatric Inventory (NPI) [behavior]
  * quality of life (QOL) -AD

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Dubois, Prof., Principal Investigator — Centre des Maladies Cognitives et Comportementales, Federation des maladies du systeme nerveux, Hoptial de la Salpetriere, Pavillon Paul Castaignes (Sous-sol), 47-83 Bd de l'Hopital, 75651 Paris Cedex 13
Locations (27):
- Austria (6):
  - Landeskrankenhaus Hall Gedächtnisambulanz, Hall in Tirol
  - LNK Wagner-Jauregg, Dept. of geriatrics, Linz
  - Christian Doppler Klinik, Univ. Klinik f. Neurologie, Salzburg
  - MUW Klin. Pharmakologie und Klinik für Neurologie, Vienna
  - MUW, Klin.Abt.f. Biolog. Psychiatrie, Vienna
  - SMZ-Ost, Psychiatric Dep., Vienna
- Croatia (4):
  - Klinčki Bolnički Centar Rijeka, Klinika za Psihijatriju, Rijeka
  - Opća bolnica Varaždin, Klinika za Neurologiju, Varaždin
  - "BONIFARM" Poliklinika za kliničku farmakologiju i toksikologiju, Zagreb
  - Psihijatrijska Bolnica Vrapče, Zagreb
- Czechia (2):
  - University Thomayer Hospital, Prague
  - University Hospital Motol, Clinic of Neurology, Prague
- France (7):
  - CMRR Hôpital Pellegrin, Bâtiment USN Tastet Girard, Bordeaux
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Centre Hospitalier Universitaire (CHU) de Dijon, Dijon
  - Centre Mémoire de Ressources et de Recherche, Service de Neurologie, Montpellier
  - Hôpital de la Pitié-Salpêtrière, Paris
  - CHU de Rennes Site Hôtel Dieu, Rennes
  - Hopital La Grave, Toulouse
- Germany (7):
  - Charite Universitätsmedizin Berlin, Klinik u. Hochschulambulanz f. Psychiatrie u. Psychotherapie, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Klinik für Psychiatrie und Psychotherapie, Hamburg
  - Arzneimittelforschung Leipzig GmbH, Studienzentrum, Leipzig
  - Zentralinstitut für Seelische Gesundheit, Abt. Gerontopsychiatrie, Mannheim
  - Klinik u. Poliklinik f. Psychiatrie u. Psychotherapie der TU München, Munich
  - Studienzentrum PD Dr. Steinwachs, Nuremberg
  - NeuroPoint GmbH, Ulm/Donau
- EPAMED, s.r.o., Košice, Slovakia